CLINICAL TRIAL: NCT06383715
Title: Acceptability and Feasibility of a Congitive Behavioral Therapy Workshop for Content Moderators: a Pilot Study
Brief Title: Congitive Behavioral Therapy Workshop for Content Moderators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Valencia (Other)
Responsible Party: Principal Investigator, Carlos López-Pinar, Lecturer and Researcher, Universidad Europea de Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-624
Record Dates: First submitted 2024-04-16; First posted 2024-04-25 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Work-Related Condition; Work-Related Stress Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive Behavioural Workshop (Experimental): The experimental group will attend 4 weekly group sessions of 90 minutes each. The intervention will be delivered by a Ph.D. clinical psychologist with over 15 years of clinical experience.
  Interventions: Behavioral: Cognitive-Behavioral Therapy Workshop for Content Moderators

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy Workshop for Content Moderators — This 4-session group workshop is based on the principles of Cognitive Behavioral Therapy. It consists of four sessions:
  1. Presentation. Scientific evidence of psychological consequences on content moderatos. Psicoeducation on the effects of vicarious trauma exposure.
  2. Presentation of the cognitive model. Identification/operationalization of thoughts. Discussion of possible irrational thoughts.
  3. Psychoeducation of emotions and their adaptive function. Behavioral strategies of emotions: exposure therapies and behavioral activation.
  4. The role of social support. Strategies for appropriate work and sleep hygiene. Strategies for maintaining gains. Farewell.

SUMMARY:
Professional content moderators play a critical role in preventing Internet users from being exposed to more sensitive content. However, recent literature has shown that this work places content moderators at increased risk for several psychological outcomes, including intrusive thoughts and vicarious stress trauma. This pilot study will assess the acceptability and feasibility of a brief (4-session) cognitive-behavioral workshop to reduce these risks.

DETAILED DESCRIPTION:
The growing amount of user-generated content is forcing companies to hire more and more content moderators (CMs). There is ample empirical evidence that exposure to the trauma of others at work affects well-being and mental health , and research focused on CMs suggests that they experience similar effects as other professionals. This includes an increased risk of developing syndromes such as secondary posttraumatic stress, vicarious trauma, and burnout. Recent literature, although limited, indicates that CMs are already using coping strategies such as creating boundaries between work and personal life, although they expressed a preference for individual therapy with specialized professionals. However, this initial work points to the need for technology companies to develop prevention programs based on preventing exposure to traumatic content (.

Therefore, a CBT workshop consisting of four 90-minute group sessions was designed specifically to prevent work-related consequences in a small sample of content moderators. The workshop will have a cognitive-behavioral orientation, which has been shown to be more effective for posttraumatic symptoms. Psychological distress, PTSD symptoms, job satisfaction, and coping strategies will be measured before and after the intervention to assess the feasibility of the workshop.

ELIGIBILITY:
Inclusion Criteria:

* Actively work as a professional content moderator, for at least 6 months.

Exclusion Criteria:

* Presence of a psychotic or personality disorder as defined by DSM-5 criteria.
* Receive another psychological treatment during the time of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
The Kessler Psychological Distress Scale (K10) | Week 0, week 4, and week 12
  It is a simple measure of psychological distress. The K10 scale involves 10 questions about emotional states each with a five-level response scale. The measure can be used as a brief screen to identify levels of distress. The tool can be given to patients to complete, or alternatively the questions can be read to the patient by the practitioner.

SECONDARY OUTCOMES:
Work Satisfaction Scale, JobStat'73 | Week 0, week 4, and week 12
  It is made up of 5 questions related to their satisfaction with the job, possible continuity in it and whether they would recommend it to others.
Coping Mechanisms Scale | Week 0, week 4, and week 12
  It measures how the participant cope with stress, collecting data from 16 strategies.
PTSD Checklist-Civilian Version (PCL-C) | Week 0, week 4, and week 12
  The PCL-C includes 17 items assessing a variety of symp- tomatic responses to stress, and respondents self-reported the extent to which they were bothered by these symptoms, within the past month, on a scale from 1 (Not at all) to 5 (Extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos López-Pinar, PhD, Principal Investigator — Universidad Europea de Valencia
Locations (1):
- MEGA cloud services, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Léonard, M.-J., Saumier, D., & Brunet, A. (2020). When the lawyer becomes traumatized: A scoping review. SAGE Open, 10(3), 1-10. https://doi.org/10.1177/2158244020957032
- [Background] Lewis C, Roberts NP, Andrew M, Starling E, Bisson JI. Psychological therapies for post-traumatic stress disorder in adults: systematic review and meta-analysis. Eur J Psychotraumatol. 2020 Mar 10;11(1):1729633. doi: 10.1080/20008198.2020.1729633. eCollection 2020. PMID 32284821
- [Background] Seigfried-Spellar, K. C. (2018) Assessing the Psychological Well-being and Coping Mechanisms of Law Enforcement Investigators vs. Digital Forensic Examiners of Child Pornography Investigations. Journal of Police and Criminal Psychology, 33, 215-226. https://doi.org/10.1007/s11896-017-9248-7
- [Background] Steiger, M., Bharucha, T. J., Venkatagiri, S., Riedl, M. J., & Lease, M. (2021). The psychological well-being of content moderators: The emotional labor of commercial moderation and avenues for improving support. In CHI '21: Proceedings of the 2021 CHI Conference on Human Factors in Computing Systems (pp. 1-14). ACM. https://doi.org/10.1145/3411764.3445092
- [Background] Spence, R., Bifulco, A., Bradbury, P., Martellozzo, E., & DeMarco, J. (2023a). The psychological impacts of content moderation on content moderators: A qualitative study. Cyberpsychology: Journal of Psychosocial Research on Cyberspace, 17(4), Article X. https://doi.org/10.5817/CP2023-X-X